CLINICAL TRIAL: NCT06198205
Title: Effects of Fundamental Motor Skills Program on Motor and Cognitive Abilities in School Going Children
Brief Title: Effects of Fundamental Motor Skills Program on Motor and Cognitive Abilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0755
Record Dates: First submitted 2023-12-26; First posted 2024-01-10 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Child Development
Keywords: Cognition.; Fundamental motor skills; School going children

STUDY DESIGN:
Intervention Model Description: it is a randomized control trial, used to compare Effects of Fundamental Motor Skills Program on Motor and Cognitive Abilities in school going children. Subjects meeting the predetermined inclusion and exclusion criteria will be divided into two groups using simple random sampling technique.
Who Masked: Participant
Masking Description: participants will get separate treatment protocols and possible efforts will be put to mask the both groups about their treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Students will participate in fundamental motor skills(FMS) program that will include 12 basic motor skills.
  Interventions: Other: Fundamental motor skills
- Group B (Experimental): Group B students will do their regular afterschool programs unstructured child's free play
  Interventions: Other: Regular after school program

INTERVENTIONS:
Other: Fundamental motor skills — This will receive fundamental motor skills(FMS) program include 12 basic motor skills(running,hopping,galloping,leaping,jumping,sliding,strinking,dribbling,catching overhand throwing and underhand rolling)
  Arms: Group A
Other: Regular after school program — This group will receive regular afterschool programs unstructured child's free play which include sliding, hide and seek, sea-saw, and running along with reading, drawing. Each intervention session lasted 60 minutes. The study will be conducted in the duration of 8 weeks with 3 sessions per week (total 24 sessions) will be given to the students.
  Arms: Group B

SUMMARY:
School age child development is a range from 6 to 12 years of age. During this time period observable differences in height, weight, and build of children may be prominent. The language skills of children continue to grow and many behavior changes occur as they try to find their place among their peers. School-age children gain between four and seven pounds each year., Increases in height will vary, and a three-to-six height difference in age groups is typical. Growth spurts are common in school-age children, as are periods of slow growth. Fundamental Movement Skills (FMS) are a specific set of gross motor skills that involve different body parts. These skills are the building blocks for more complex skills that children will learn throughout their lives. They help children take part in games, sports and recreational activities. While the Motor cognition takes into account the preparation and production of actions, as well as the processes involved in recognizing, predicting, mimicking, and understanding the behavior of other people It will be a randomized controlled trial. This study will include 48 school going children who meet the inclusion criteria will be recruited from Qazi Grammer School, The Cardour School. Two groups will be formed and 24 students will be allocated in each group. Before applying the techniques pre and post reading will be taken.Tools used during our study will be Parent proxy report format and Six minutes Walk test and portage guide to early education. In Group A which will be experimental group Experimental Group students will participate in fundamental motor skills(FMS) program that will include 12 basic motor skills(running,hopping,galloping,leaping,jumping,sliding,strinking,dribbling,catching overhand throwing and underhand rolling) will be applied and Group B which will be control group regular afterschool programs which include unstructured child's free play including sliding, hide and seek, sea-saw, and runing, along with reading, drawing will be used. These activities will continue for 3 sessions per week for the period of 8 weeks. Data will be analyzed by using SPSS for windows version 25.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial, used to compare the effects of Effects of Fundamental Motor Skills Program on Motor and Cognitive Abilities in school going children.

Subjects meeting the predetermined inclusion and exclusion criteria will be divided into two groups using simple random sampling technique. Assessment will be done by using The Portage Guide to Early Education, Six minutes Walk test and PEDsQL Parent proxy report format. Subjects in group A will be participated in fundamental motor skills(FMS) program and subjects in group B will be participated in regular after school programs unstructured child's free play.

ELIGIBILITY:
Inclusion Criteria:

* • Age: school going children of age between 5 to 6 years.

  * Students who are present at school in their afterschool programs between 12 to 2pm.
  * Gender: both boys and girls.
  * Children who are physically active
  * Children who are able to understand command
  * BMI= Normal to Obese(16.5 - >28.0).

Exclusion Criteria:

* Students with any leg length discrepancy .
* With any surgical intervention from last 6 months
* Any history of fracture.
* Children with flat foot/club foot.
* Children with genu varum/valgum

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
The Portage Guide to Early Education | duration of 8 weeks with 3 sessions per week(total 24 sessions)
  The Portage Guide to Early Education is a develop- mentally formulated curriculum to be used with children, either handicapped or normal, between the mental ages of birth to five years. Maximum value of portage guide to early education showed the improvement of the training increased value showed improved motor and cognitive abilities of the patient. Each question's answer of motor and cognitive part of the portage guide to early education was calculated by the formula, Correct answer÷ incorrect answer× 12...then add all the answers of both components and divided it by 2,we divided it by two because in our study we include only two components of this questionnaire instead of all 5
Six minutes Walk test | duration of 8 weeks with 3 sessions per week(total 24 sessions)
  In healthy children, the 6-min walk test is a reliable and valid functional test for assessing exercise tolerance and endurance. An individual's response to exercise is an important clinical assessment tool, since it provides a composite assessment of their respiratory, cardiac and metabolic systems. The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance.
PEDsQL Parent proxy report format | duration of 8 weeks with 3 sessions per week(total 24 sessions)
  Parent proxy-report includes ages 2-4 (toddler), 5-7 (young child), 8-12 (child), and 13-18 (adolescent), and assesses parent's perceptions of their child's HRQOL. The items for each of the forms are essentially identical, differing in developmentally appropriate language, or first or third person tense. The PedsQL achieved excellent reliability across scales, and distinguished healthy individuals from those with chronic health conditions, as well as individuals with ASD from those without. Factor analysis confirmed a 5-factor model.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Asif Javed, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia-Hermoso A, Alonso-Martinez AM, Ramirez-Velez R, Perez-Sousa MA, Ramirez-Campillo R, Izquierdo M. Association of Physical Education With Improvement of Health-Related Physical Fitness Outcomes and Fundamental Motor Skills Among Youths: A Systematic Review and Meta-analysis. JAMA Pediatr. 2020 Jun 1;174(6):e200223. doi: 10.1001/jamapediatrics.2020.0223. Epub 2020 Jun 1. PMID 32250414